CLINICAL TRIAL: NCT07347119
Title: Prospective Geometric Analysis of Ultra-Widefield OCTA Characteristics in Central Serous Chorioretinopathy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Director of ophthalmology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Other Study IDs: 2025KYPJ135
Record Dates: First submitted 2025-12-17; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Central Serous Chorioretinopathy (CSC)
Keywords: Central Serous Chorioretinopathy; Ultra-Widefield Optical Coherence Tomography Angiography; Geometry
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Central Serous Chorioretinopathy: Clinically, serous retinal detachment (SRD) can be detected via fundus examination and optical coherence tomography (OCT), along with focal or multifocal retinal pigment epithelium (RPE) changes confined to small pigment epithelial detachment (PED) lesions. Fundus fluorescein angiography (FFA) demonstrates RPE leakage. SRD typically resolves within 3-4 months, and in most cases, no long-term symptoms persist except for color discrimination deficits in some patients.
- Chronic Central Serous Chorioretinopathy: When the disease course exceeds 4-6 months, obvious multifocal atrophic retinal pigment epithelium (RPE) changes, multifocal leakage, and extensive RPE atrophy can be observed. Fundus autofluorescence (FAF) shows hypofluorescence in the RPE-damaged areas.
- Recurrent Central Serous Chorioretinopathy: The patient has a history of one or more previous episodes, during which the symptoms completely resolved or significantly improved, and optical coherence tomography (OCT) examination showed complete absorption of subretinal fluid, with reattachment of the neurosensory retina. After complete remission of the first (or previous) episode (an interval of at least 3-6 months is generally considered), the patient develops typical symptoms of central serous chorioretinopathy (CSC) again, accompanied by objective evidence of the acute or chronic phase, such as changes detected by OCT or fundus fluorescein angiography (FFA).
- Control Group: Healthy control subjects without any local or systemic diseases

SUMMARY:
By leveraging parameters including fractal dimension and topological index, we constructed a quantitative evaluation framework for ultra-widefield optical coherence tomography angiography (UWF-OCTA) images in patients with central serous chorioretinopathy (CSC), thus overcoming the limitations of conventional qualitative analysis.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is a macular disorder characterized by choroidal hyperpermeability and serous retinal detachment, with chronicity leading to irreversible visual impairment. Optical coherence tomography angiography (OCTA) allows non-invasive, high-resolution 3D imaging of choroidal microcirculation, but traditional OCTA analysis relies on qualitative assessment, which cannot quantify vascular structural heterogeneity.

This prospective cohort study will enroll 120 subjects, including CSC patients and healthy controls, who will be allocated to acute, chronic, recurrent CSC groups, or healthy control group. Ultra-widefield swept-source OCTA (UWF SS-OCTA) will be used to capture choroidal vascular images. Geometric parameters (fractal dimension, topological index, 3D vascular diameter) will quantify vascular complexity, distribution, and morphology. Strict inclusion/exclusion criteria and matching for age, gender, and refraction will ensure baseline comparability. Follow-up visits will be conducted at 1, 3, 6, and 12 months post-treatment, with repeated OCTA to evaluate dynamic changes in geometric parameters and their associations with treatment response.

This study innovatively integrates geometric methods with UWF-OCTA to establish a quantitative choroidal vascular evaluation framework for CSC. It aims to identify stage-specific vascular characteristics, explore correlations between geometric markers (e.g., dynamic fractal dimension changes) and the efficacy of laser photocoagulation/anti-VEGF therapy, and validate these markers as non-invasive prognostic indicators. UWF-OCTA will enable comprehensive detection of vascular abnormalities, providing evidence for precise CSC management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years, inclusive;
* Clinical diagnosis of central serous chorioretinopathy (CSC);
* Completion of fundus fluorescein angiography (FFA) and indocyanine green angiography (ICGA) examinations;
* Completion of ultra-widefield optical coherence tomography angiography (UWF-OCTA) imaging;
* No prior history of pharmacological or surgical treatment for CSC;
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

-Presence of other ophthalmic diseases that may affect retinal or choroidal imaging or analysis, including but not limited to: Significant refractive media opacities interfering with OCTA imaging (e.g., severe cataract, vitreous hemorrhage);

* Presence of systemic diseases that may affect study outcomes or participant safety;
* Pregnant or lactating women;
* History of psychiatric or mental disorders that may impair compliance;
* Hemorrhagic diathesis or requirement for long-term anticoagulant therapy;
* History of long-term systemic medication use that may affect choroidal or retinal circulation;
* Presence of severe and/or uncontrolled comorbid medical conditions, including but not limited to:

Uncontrolled diabetes mellitus; Uncontrolled hypertension; Active uncontrolled infection; Chronic obstructive pulmonary disease (COPD) with dyspnea at rest;

* History of intraocular surgery or intravitreal injection within the past 6 months;
* High refractive error defined as:

Spherical equivalent (SE) < -6.0 diopters or > +3.0 diopters, or Axial length (AL) > 26.0 mm;

-Any other condition that, in the opinion of the investigator, would make participation unsafe or interfere with protocol adherence.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study subjects were recruited from outpatients of the Medical Retina Department at Zhongshan Ophthalmic Center, and eligible cases meeting the study criteria were selected from the outpatient medical record system.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Choroidal Vascular Fractal Dimension | Baseline, 1 month, 3 months, 6 months, and 12 months
  Choroidal vascular fractal dimension quantified from optical coherence tomography angiography (OCTA) images.

SECONDARY OUTCOMES:
Maximum subretinal fluid height | Baseline, 1 month, 3 months, 6 months, and 12 months
  The maximum height of subretinal fluid measured in micrometers (μm) on optical coherence tomography angiography (OCTA) images.
Subretinal fluid area | Baseline, 1 month, 3 months, 6 months, and 12 months
  The basal area of subretinal fluid measured in square millimeters (mm²) on optical coherence tomography angiography (OCTA) images.
Subretinal fluid volume | Baseline, 1 month, 3 months, 6 months, and 12 months
  The volume of subretinal fluid measured in cubic millimeters (mm³) on optical coherence tomography angiography (OCTA) images.
Choroidal vascular branching index | Baseline, 1 month, 3 months, 6 months, and 12 months
  The branching index of choroidal blood vessels quantified from optical coherence tomography angiography (OCTA) images.
Choroidal Vascular Connectivity Index | Baseline, 1 month, 3 months, 6 months, and 12 months
  The connectivity index of choroidal blood vessels quantified from optical coherence tomography angiography (OCTA) images.
Mean curvature of choroidal blood vessels | Baseline, 1 month, 3 months, 6 months, and 12 months
  The mean curvature of choroidal blood vessels quantified from optical coherence tomography angiography (OCTA) images.
Mean curvature of retinal blood vessels | Baseline, 1 month, 3 months, 6 months, and 12 months
  The mean curvature of retinal blood vessels quantified from optical coherence tomography angiography (OCTA) images.

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, PH.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong 510060
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided